CLINICAL TRIAL: NCT06183736
Title: A Single-arm, Open-label, Multicenter, Phase II Study of CVL237 Tablets in the Treatment of Advanced Solid Tumors With PTEN Deficiency
Brief Title: CVL237 Tablets in the Treatment of Advanced Solid Tumors With PTEN Deficiency
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Convalife (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVL237-P2001
Record Dates: First submitted 2023-11-26; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Advanced Solid Tumors
Keywords: PTEN deficiency; gastric cancer; prostate cancer; endometrial cancer; colorectal cancer; lung cancer; breast cancer; melanoma; CVL237 Tablets
MeSH Terms: conditions — Stomach Neoplasms; Prostatic Neoplasms; Endometrial Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Breast Neoplasms; Melanoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single-arm (Experimental): This is a single-arm, open-label, multicenter, phase II study of CVL237 tablets in the treatment of advanced solid tumors with PTEN deficiency.All patients will be given CVL237 tablets, 200 mg, taken with food once daily for 28 consecutive days as a treatment cycle.
  Interventions: Drug: CVL237 tablets

INTERVENTIONS:
Drug: CVL237 tablets — CVL237 tablets, 200 mg, taken with food once daily for 28 consecutive days as a treatment cycle.

SUMMARY:
This is a single-arm, open-label, multicenter, phase II study of CVL237 tablets in the treatment of advanced solid tumors with PTEN deficiency. It is planned to enroll patients with PTEN deficiency advanced solid tumors of different tumor types (PTEN deficiency gastric cancer, prostate cancer, endometrial cancer, colorectal cancer, lung cancer, breast cancer and melanoma etc.) to evaluate the preliminary efficacy, safety and pharmacokinetic profile of CVL237 tablets in patients with PTEN deficiency advanced solid tumors of different tumor types.

DETAILED DESCRIPTION:
"The predicted BSC (best supportive care treatment) ORR is 0.5% and the post-treatment ORR is 15% with 80% certainty and a significance level of 0.05 (bilateral). The first stage: After testing the drug on 10 patients in the first stage, the trial will be terminated if 0 respond; if any subject showed respond then enter the second stage; The second stage: If the trial goes on to the second stage, another 4 evaluation subjects could continue to be enrolled, a total of 14 patients will be studied. If the total number responding is less than or equal to 0, the drug is rejected.. If a subject falls off during the trial, i.e., the objective remission cannot be judged, the number of subjects should be completed.

The maximum number of qualified subjects for the 7 tumor types is 98 (in the best case, according to clinical practice, it is recommended to enroll a certain number of subjects for each tumor type, not exceeding 14).

CVL237 tablets, 200 mg, taken with food once daily for 28 consecutive days as a treatment cycle.

Tumors will be evaluated according to the Solid Tumor Efficacy Evaluation Criteria (RECIST version 1.1 criteria) and will be assessed every 2 cycles. Tumor assessment may be increased by the investigator as clinically indicated. Treatment periods may be administered continuously until the onset of intolerable adverse effects, disease progression, withdrawal of informed consent (ICF), lost to follow-up, death, or study termination, whichever occurs earliest. Efficacy of each tumor type will be analyzed independently.

Withdrawal from the study/termination of treatment for any reason required return to the study center for safety follow-up 30 days (±3 days) after the last dose. Patients will then enter a survival follow-up period until the full 2 years after the end of the trial/missing/death. All patients will be followed up every 12 weeks (±5 days) for survival, either by telephone with the subject, their family or local hospital.

Pharmacokinetic studies will be performed in 6-12 patients."

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years (including those of 18 and 75 years old; patients over 60 years old cannot have more than 3 kinds of complications of heart, lung, liver and kidney function at the same time); the sex is not limited;
2. Aged 18-75 years (including those of 18 and 75 years old; patients over 60 years old cannot have more than 3 kinds of complications of heart, lung, liver and kidney function at the same time); the sex is not limited;after standard treatment as determined by the investigator, or for whom there is no standard treatment, or who refuse the standard treatment;
3. PTEN deficiency will be determined based on analysis of patient tumor samples and by testing PTEN protein expression using immunohistochemistry (IHC) at the central laboratory;
4. Have at least one measurable lesion that meets the requirements of RECIST 1.1 ; If the lesion previously treated with local therapy (radiotherapy, ablation, interventional therapy, etc.) is the only lesion, there must be unequivocal imaging evidence of disease progression in this lesion;
5. Eastern Cooperative Oncology Group (ECOG) score: 0-2;
6. Expected survival time of more than 3 months;
7. Good organ function level:

   * Absolute neutrophil count (ANC)≥ 1.5 × 10^9/L
   * Platelets (PLT)≥ 75 × 10^9/L
   * Hemoglobin (Hb)≥ 90 g/L
   * Total bilirubin (TBIL)≤ 1.5 × ULN
   * Alanine aminotransferase (ALT)≤ 2.5 × ULN;Patients with liver metastases or liver cancer: ≤ 5 × ULN
   * Aspartate aminotransferase (AST)≤ 2.5 × ULN;Patients with liver metastases or liver cancer: ≤ 5 × ULN
   * Serum creatinine clearance (Ccl)≤ 1.5 × ULN, or ≥ 60 mL/min (calculated according to the Cockcroft-Gault formula)
   * Activated partial thromboplastin time (APTT)≤ 1.5 × ULN
   * International Normalized Ratio (INR)≤ 1.5 × ULN
   * Ejection fraction (LVEF) ≥ 50% and Fridericia-corrected QT interval (QTcF) < 450 ms for males and < 470 ms for females
8. Eligible patients (males and females) of childbearing potential must agree to use a reliable method of contraception (hormonal or barrier method or abstinence) with their partner during the study and for at least 180 days after the last dose; Females of childbearing potential must not be breastfeeding, and females of childbearing potential must have a negative pregnancy test before the start of dosing;
9. Voluntarily participate in this clinical trial, understand the study procedures and be able to sign the ICF in writing.

Exclusion Criteria:

1. Patients who have progressed on previous treatment with any PI3K, mTOR or AKT inhibitors (except for patients who dropped out due to intolerance);
2. Known hypersensitivity to any ingredient of CVL237;
3. Those requiring OATP1B1 and OATP1B3 substrate drugs, CYP3A4/5 substrate drugs, moderate and potent cytochrome P450 3A4/5 inhibitors, and potent inducers of cytochrome P450 3A4/5 for treatment;
4. Received chemotherapy, radiotherapy, immunotherapy, biological agents, molecular targeted therapy or endocrine therapy and other antitumor drugs within 4 weeks before the first dose of the study drug, except for the following: nitrosoureas or mitomycin C within 6 weeks before the first dose of the study drug; oral fluorouracils and small molecular targeted drugs within 2 weeks before the first dose of the study drug or 5 half-lives of the drug (whichever is shorter);
5. Participated as a subject in a clinical trial within 4 weeks prior to the first dose of the study drug;
6. Patients who have undergone major organ surgery (excluding needle biopsy) or significant trauma within 4 weeks prior to the first dose of the study drug, or require selective surgery during the study;
7. Previously received allogeneic bone marrow transplantation or solid organ transplantation;
8. Presence of third space fluid accumulation (such as massive pleural effusion and ascites) that cannot be controlled by drainage or other methods;
9. The adverse reactions to previous antitumor treatment have not recovered to CTCAE 5.0 grade ≤ 1 (except for alopecia and other toxicities judged by the investigator to have no safety risk);
10. Patients with active brain metastasis, meningeal metastasis and central nervous system (CNS) involvement, who are not suitable for enrollment as judged by the investigator;
11. Participants with impairment of gastrointestinal (GI) function or GI disease that, in the judgment of the investigator, could significantly alter the absorption of the study drug (e.g., ulcerative disease, uncontrollable nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection);
12. Subjects with a history of acute pancreatitis within 1 year prior to screening or subjects with a previous history of chronic pancreatitis;
13. Uncontrolled pulmonary fibrosis, acute lung disease, interstitial lung disease, FEV1 (post-bronchiectasis) < 70% predicted value at screening, or hepatic failure, etc.;
14. Patients with active viral, bacterial, fungal or other infections requiring systemic treatment (such as active pulmonary tuberculosis), excluding nail bed fungal infection;
15. Patients with HBV or HCV infection (defined as HbsAg and/or HbcAb positive and HBV DNA copies ≥ 1 × 104 copies/mL or ≥ 2000 IU/mL) or acute or chronic active hepatitis C;
16. Patients with a history of immune deficiency, including positive HIV test, or other acquired or congenital immune deficiency diseases, or a history of organ transplantation, allogeneic bone marrow transplantation, or autologous hematopoietic stem cell transplantation;
17. Had any heart disease within 6 months, including: (1) Angina pectoris; (2) Arrhythmia that requires medication or is clinically significant; (3) Myocardial infarction; (4) Cardiac failure; (5) Patients with any other heart disease judged by the investigator to be unsuitable for this study;
18. Other concomitant diseases that seriously jeopardize the safety of the patient or affect the completion of the study [e.g. Uncontrolled hypertension (systolic/diastolic blood pressure ≥ 140/90 mmHg after administration of antihypertensive drugs), diabetes mellitus (HbA1c ≥ 8.0% (63.9 mmol/mol), thyroid disease, etc.] according to the judgment of the investigator;
19. Received a live vaccine within 30 days prior to the first dose of the study drug, or plan to receive a live vaccine during the study;
20. The investigator considers that there are other reasons for the unsuitability of the subject participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) in patients with PTEN deficiency as assessed according to RECIST v1.1 | Throughout the study for approximately 2 years
  objective response rate (ORR), which refers to the proportion of patients whose tumor shrinkage reaches a certain amount and maintains for a certain time, including complete response (CR) and partial response (PR)

SECONDARY OUTCOMES:
Duration of response (DOR) | Throughout the study for approximately 2 years
  Duration of response (DOR),defined as the time from the first tumor assessment of CR or PR to the first tumor assessment of PD or death due to any cause.
Disease control rate (DCR) | Throughout the study for approximately 2 years
  Disease control rate (DCR),which refers to the proportion of patients whose tumors shrink or remain stable for a certain time (mainly for solid tumors), including CR, PR and SD
Progression-free survival (PFS) | Throughout the study for approximately 2 years
  Progression-free survival (PFS), defined as the time from the start of study treatment to any documented tumor progression or death due to any cause, whichever occurs first;
Overall survival (OS) | Throughout the study for approximately 2 years
  Overall survival (OS), defined as the time from enrollment to death due to any cause. Efficacy of each tumor type will be analyzed independently.

CONTACTS AND LOCATIONS:
Locations (1):
- Li Ning, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No